CLINICAL TRIAL: NCT01832454
Title: Safety and Efficacy of Bone Marrow MNC for the Treatment of Cerebral Palsy in Subjects Below Years. It is Self Funded (Patients' Own Funding) Clinical Trial
Brief Title: Safety and Efficacy of Bone Marrow MNC for the Treatment of Cerebral Palsy in Subjects Below 15 Years
Acronym: BMCP2
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chaitanya Hospital, Pune (Other)
Responsible Party: Principal Investigator, Dr. Sachin Jamadar, CO-Investigator, Chaitanya Hospital, Pune
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 00160
Record Dates: First submitted 2013-02-26; First posted 2013-04-16 (Estimated); Last update posted 2014-09-17 (Estimated); Status verified 2014-09

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy stem cells [MNCS]
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intra thecal inj of autologous MNC (Other): Intra thecal inj of autologous MNC
  Interventions: Other: Intra thecal inj of autologous MNC

INTERVENTIONS:
Other: Intra thecal inj of autologous MNC — Intra thecal inj of autologous MNC

SUMMARY:
This Study is Single arm, Single Centre trail to check the safety and efficacy of bone marrow derived autologous mononuclear cells(100 millions per dose )trial to be conducted for 36 months in 100 patients ( below 15 years of age) with cerebral palsy in India. Primary outcome measures are improvement in walking ability and kinetic gait pattern.

DETAILED DESCRIPTION:
This Study is Single arm, Single Centre trail to check the safety and efficacy of bone marrow derived autologous mononuclear cells(100 millions per dose )trial to be conducted for 36 months in 100 patients ( below 15 years of age) with cerebral palsy in India. Primary outcome measures are improvement in walking ability and kinetic gait pattern

ELIGIBILITY:
Inclusion Criteria:

* Subject aged above 3 years and below 15 years with a diagnosis of Cerebral Palsy.
* Regional Nerve damage as shown by Magnetic Resonance Imaging(MRI)
* Able to Comprehend and give written informed consent form for the study
* willing to come to the hospital for follow up visits as per the protocol requirements

Exclusion Criteria:

* History of meningitis,meningoencephalits,epilepsy or life threatening allergic or immune -mediated reaction 2
* Hemodynamically unstable patients
* history of or concurrent autoimmune disease or acute episode if Guillain- barre syndrome
* peripheral Muscular dystropy

Ages: 3 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2011-03; Primary Completion 2015-11 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Improvement in muscle rigidity using Ash worth scale and overall motor control using oxford scale. | 6 months
  - Improvement in muscle rigidity using Ash worth scale and overall motor control using oxford scale at Time point - 6 Months.

SECONDARY OUTCOMES:
-Improvement in IQ by using Benit Kamat scale. | 6 Months
  -Improvement in IQ by using Benit Kamat scale. Improvement in social behaviour. Reduction in deformity.

CONTACTS AND LOCATIONS:
Overall Officials: Anant E Bagul, M.S., Principal Investigator — chaitanya stem cell centre
Locations (1):
- Chaitnany Hospital, Pune, Maharashtra, India